CLINICAL TRIAL: NCT07014410
Title: A Multicenter Phase II Clinical Study of Pyrotinib Combined With Dalpiciclib Combined With Letrozole in the Treatment of ER-positive and HER2-positive Advanced Breast Cancer
Brief Title: Pyrotinib Combined With Dalpiciclib Combined With Letrozole in ER-positive and HER2-positive Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Zhanhong, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPYLET
Record Dates: First submitted 2023-05-05; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pyrotinib dalpiciclib letrozole (Experimental): Patients receive pyrotinib 320mg/d, dalpiciclib 125mg/d and letrozole 2.5mg/d until disease progression, intolerated toxicity.
  Interventions: Drug: pyrotinib dalpiciclib letrozole

INTERVENTIONS:
Drug: pyrotinib dalpiciclib letrozole — ER positive HER2 positive advanced breast cancer patients are given pyrotinib+dalpiciclib+letrozole
  Other Names: Femar

SUMMARY:
This is a a multicenter Phase II clinical study investigating efficacy of pyrotinib combined with dalpiciclib combined with letrozole in ER-positive and HER2-positive advanced breast cancer patients. The sample size is 63.

DETAILED DESCRIPTION:
This is a a multicenter Phase II clinical study investigating efficacy of pyrotinib combined with dalpiciclib combined with letrozole in ER-positive and HER2-positive advanced breast cancer patients. Patients receive pyrotinib 320mg/d, dalpiciclib 125mg/d, d1-21, q28d. One cycle is 28d.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study, signed the informed consent, and had good compliance
2. Postmenopausal or premenopausal/perimenopausal women aged ≥18 years and ≤75 years
3. Patients with recurrent/metastatic breast cancer confirmed by histopathology with positive ER expression and positive HER2 expression
4. Have at least one extracranial measurable lesion that meets RECIST 1.1 criteria
5. At most one previous trastuzumab containing systemic therapy for recurrent metastatic breast cancer

Exclusion Criteria:

1. Subjects had untreated central nervous system metastasis
2. Bilateral breast cancer, inflammatory breast cancer, or latent breast cancer
3. Previous treatment with any CDK4/6 inhibitors
4. Inability to swallow, intestinal obstruction, or other factors affecting drug use and absorption
5. Subject has had other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within 5 years or at the same time

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | through study completion, an average of 2 year
  the proportion of patients achieving complete response or partial response

SECONDARY OUTCOMES:
Progression Free Survival | through study completion, an average of 2 year
  Time to progression or death, which comes first

CONTACTS AND LOCATIONS:
Overall Officials: Zhanhong Chen, Master, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No